CLINICAL TRIAL: NCT02749838
Title: Characterization of Human Cancers by Molecular Profiling of Patient Biospecimens
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Pharmatech (Industry)
Collaborators: Paradigm (Unknown)
Responsible Party: Sponsor
Other Study IDs: PI-13-1008
Record Dates: First submitted 2014-06-02; First posted 2016-04-25 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Cancer
Keywords: Cancer; Genomic testing; Genetic testing; Molecular screening; Molecular Profiling; Biomarker; Biopsy; Tumor sampling; Registry
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
Purpose of the Protocol:

* To prospectively identify cancer patients whose tumors express specific molecular markers targeted by therapeutic agents, for the purpose of selecting the most clinically appropriate anticancer therapy, including clinical trial opportunities.
* To collect and analyze biospecimens from cancer patients, using primarily standard of care laboratory methods, for the purpose of determining the expression of specific genotypic and phenotypic disease markers of scientific and medical interest.
* To create a protocol database, including case and disease stage-matched clinical and therapeutic history data in addition to patient biomarker profiles, to serve as:

  * a systematic collection of data for comparing patient data to clinical trial selection criteria for the purpose of informing a clinical investigative site of available clinical trials matching patient clinical status;
  * a collection of clinically matched, comprehensive molecular results for scientific and research and development applications.

DETAILED DESCRIPTION:
The molecular understanding of cancer is advancing rapidly, and a new generation of more effective, targeted cancer drugs are taking center stage in cancer care. Yet the investigators system for clinical testing of new agents has not kept pace with the revolution in cancer biology.

Stratification by genotypic and phenotypic abnormalities further divides histological cancers into a myriad of clinically distinct subtypes. As cancer therapies become more selective, and the intent to treat populations and the predictability of patient presentation decrease, clinical trial enrollment becomes more difficult by traditional methods. A breakout solution is needed in clinical research methodology, to create a more efficient means of developing new cancer drugs in the US. Improved methods for the systematic, prospective screening of cancer patients are needed to identify the subsets of patients whose tumors express molecular markers targeted by precision therapeutics. This protocol will evaluate clinical samples of cancer tissue to identify the molecular abnormalities present in individual patients' cancer. In this context the investigators objective will be to enable physicians to more thoroughly characterize the molecular abnormalities underlying cancer and to connect eligible patients to precision treatments as part of optimal care.

By making trials more accessible and utilizing technology wisely, it should be possible to match cancer patients to appropriate treatments, including clinical trials, within a clinically relevant timeframe to bring research opportunities into consideration for best clinical care.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have given informed consent in accordance with the methods and procedures of this study
2. Diagnosis of cancer requiring medical care
3. Age ≥18 years
4. Patients under oncology care of a participating site
5. ECOG performance status of 0-3
6. Sufficient clinical status for collection of biospecimen samples within usual care

Exclusion Criteria:

1. Patients considered minors in the jurisdiction where the protocol is conducted
2. Patients who are prisoners
3. Patients who are employees of the research site
4. Relatives of the principal investigator or any participating physician
5. Patients with decisional incapacity who cannot understand or comprehend the informed consent form and therefore cannot give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There are no restrictions on number, gender, or racial/ethnic orgin of patients enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2014-05; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Identification of oncogenic molecular abnormalities by laboratory testing of tumor tissue | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthew B Wiener, PharmD, Principal Investigator — Pharmatech Inc.
Locations (1):
- Pharmatech Inc., Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No